CLINICAL TRIAL: NCT02243410
Title: Visual Analogue Scale (VAS) - a Quality Assurance Research Study to Assess the Quality of the VAS as a Means for Measuring Postoperative Pain.
Brief Title: Visual Analogue Scale - a Quality Assurance Study
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jacob Rosenberg, Professor, Herlev Hospital
Other Study IDs: HBK01
Record Dates: First submitted 2014-09-09; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It has come to our attention that there is not a general consensus of how to apply Visual Analogue Scale (VAS) as a tool in measuring pain amongst postoperative patients in Denmark.

The assumption is that patients will grade the level of pain differently dependent on how VAS is presented.

DETAILED DESCRIPTION:
To ensure the data is valid for the study it has been decided to base the research material on four different VAS usage, as it is most often used in clinical practise in Denmark. Which in this case implies VAS horizontal, with and without endpoint, and VAS vertical, with and without endpoint. Every participant will grade their pain on each of the listed VAS representations. Furthermore, as a guideline, the participant will be asked to grade the pain on a Numerical Ranking Scale (NRS).

The ordering of VAS lines will be subject to randomization, for each participant

ELIGIBILITY:
Inclusion Criteria:

* Patient must have undergone surgery within the last five days
* The patient must be able and willing to participate in the study
* Must be at 18 years of age or older
* A patient can only participate one time.

Exclusion Criteria:

* Previously included patients
* Medically treated patients Linguistic difficulties
* Mentally or physically exhausted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be postoperative patients of Department of Surgery, Department of Gynecology and Department of Orthopaedic Surgery, all based at Herlev Hospital.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
agreement in VAS values with horizontal vs vertical and with and without stop lines | First five days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, MD, Study Chair — Professor
Locations (1):
- Herlev Hospital, Herlev, Herlev, Denmark